CLINICAL TRIAL: NCT02808104
Title: A Double-Blind Placebo-Controlled Phase II Study to Determine the Efficacy, Safety, Tolerability and Pharmacokinetics of a Controlled Release (CR) Formulation of Mazindol in Adults With DSM-5 Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Mazindol Controlled Release in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NLS Pharmaceutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLS-1001
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Mazindol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mazindol Controlled Release (Experimental): Mazindol controlled release taken once daily. Dosage starting at 1 mg increasing or decreasing in increments of 1 mg depending on efficacy and tolerability. Maximum dose during the study is 3 mg taken once daily.
  Interventions: Drug: mazindol
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: mazindol

INTERVENTIONS:
Drug: mazindol

SUMMARY:
The purpose of this study is to determine whether a controlled release formulation of mazindol is more effective than a placebo in the treatment of Attention Hyperactivity Disorder (ADHD) in adults.

DETAILED DESCRIPTION:
This study is an outpatient, randomized, double-blind, placebo-controlled trial in which adult subjects with ADHD will be randomized to either oral mazindol controlled release or placebo once daily. Subjects will be treated with study medication or placebo for 6 weeks with visits occurring weekly to measure efficacy and any adverse events with adjustment of medication dosing as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a primary diagnosis of ADHD established by a comprehensive psychiatric evaluation based on DSM-5 criteria.
* Subject is functioning at an appropriate level intellectually as judged by the investigator.
* Subject has a minimum baseline score of 28 at screen and at baseline using the ADHD-RS-DSM5
* Subject has a minimum score of 4 (moderate) on the CGI-S at screening.
* Women of child-bearing potential must be non-pregnant, non-lactating, and agree to be on an acceptable method of contraception. Acceptable methods of contraception include intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable), and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
* In good general physical health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (ECG) measurement.
* Subject is fluent in written and spoken English and is willing and able to sign written informed consent prior to receipt of any study medication or beginning study procedures.
* Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

* Any primary DSM-5 Axis I disorder other than ADHD or any comorbid DSM-5 disorder that currently requires treatment.
* Lifetime history of any DSM-5 bipolar disorder
* Treatment with medications for any psychiatric or neurologic condition (e.g., amphetamines, MPH products, antidepressants, antipsychotics, mood stabilizers, anti-epileptics) or pressor agents concurrently or within 14 days of randomization.
* Concurrent medical illness that would interfere with the conduct of the study in the opinion of the investigator.
* History of significant cardiovascular disease, structural cardiac abnormality, cardiomyopathy, heart failure, serious heart rhythm abnormalities, coronary heart disease, transient ischemic attack or stroke, or other serious cardiac problems.
* Family history of sudden cardiac death.
* Clinically significant ECG abnormality or a QTc (Bazett correction) interval >450 msec.
* Resting sitting systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg.
* BMI <18 or >40 kg/m2.
* Other medications that have CNS effects on cognition or attention (e.g., sedating antihistamines or decongestants).
* Positive drug screen (UDS) at screening (with the exception of current ADHD medication).
* Concomitant use of sensitive CYPA4/5 or CYP2D6 substrates with narrow therapeutic indices.
* Pregnant or lactating.
* Ongoing psychotherapeutic treatment for the treatment of ADHD begun less than three months before entry into this study.
* Recent or current DSM-5 Substance Use Disorder of moderate or greater severity (i.e., > 4 SUD symptoms), excluding nicotine.
* Suicidal ideation within past 3 months, suicidal behavior within the past year, or a C-SSRS score of 3, 4 or 5 on ideation item.
* Evidence of any out-of-range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant by the Study Investigator.
* A history of significant drug allergy or systemic allergic disease (e.g., urticaria, atopic dermatitis), or any known/suspected hypersensitivity to any form of mazindol.
* Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Study Investigator, would make the subject unsuitable for the study or put them at additional risk.
* Treatment with an investigational drug within 30 days preceding the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale | weekly rating up to six weeks

SECONDARY OUTCOMES:
Clinical Global Improvement Scale | weekly rating up to six weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - AVIDA Clinic, Newport Beach, California
  - CNS Healthcare, Jacksonville, Florida
  - South Shore Psychiatric Services, Marshfield, Massachusetts
  - Rochester Center for Behavorial Medicine, Rochester Hills, Michigan
  - Midwest Research Group / St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Memorial Park Psychiatry / Bayou City Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wigal TL, Newcorn JH, Handal N, Wigal SB, Mulligan I, Schmith V, Konofal E. A Double-Blind, Placebo-Controlled, Phase II Study to Determine the Efficacy, Safety, Tolerability and Pharmacokinetics of a Controlled Release (CR) Formulation of Mazindol in Adults with DSM-5 Attention-Deficit/Hyperactivity Disorder (ADHD). CNS Drugs. 2018 Mar;32(3):289-301. doi: 10.1007/s40263-018-0503-y. PMID 29557078